CLINICAL TRIAL: NCT02016105
Title: A Randomized, Double-blind, Multicenter Study to Demonstrate Equivalent Efficacy and to Compare Safety and Immunogenicity of a Biosimilar Adalimumab (GP2017) and Humira® in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Study to Demonstrate Equivalent Efficacy and to Compare Safety of Biosimilar Adalimumab (GP2017) and Humira
Acronym: ADACCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP17-301; 2013-000747-11 (EudraCT Number)
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Plaque Type Psoriasis
Keywords: plaque type psoriasis; equivalent efficacy; safety and immunogenicity; GP2017; Humira®

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP2017 Adalimumab (Experimental): Study arm with intervention being studied in the protocol. Adalimumab Solution for subcutaneous injection with an initial dose of 80 mg s.c. in Week 0, followed by 40 mg s.c. eow, starting at Week 1 and ending at Week 51.
  Interventions: Drug: GP2017 Adalimumab
- Humira ® Adalimumab (Active Comparator): Humira® Adalimumab as a subcutaneous injection with an initial dose of 80 mg s.c. in Week 0, followed by 40 mg s.c. eow, starting at Week 1 and ending at Week 51.
  Interventions: Drug: Humira ® Adalimumab

INTERVENTIONS:
Drug: GP2017 Adalimumab
  Arms: GP2017 Adalimumab
Drug: Humira ® Adalimumab
  Arms: Humira ® Adalimumab

SUMMARY:
The aim of the study is to demonstrate equivalent efficacy and similarity in the safety profile of GP2017 and Humira® in patients with moderate to severe chronic plaque-type psoriasis.

DETAILED DESCRIPTION:
The aim of this study (Treatment Period 1) was to demonstrate equivalent efficacy, primarily based on the PASI75 response rate at Week 16, and similar safety of the proposed biosimilar GP2017 and Humira in patients with moderate to severe chronic plaque-type psoriasis at the end of Treatment Period 1, after 17 weeks of study treatment.

The subsequent Treatment Period 2 (Week 17 to Week 35) and the Extension Period (Week 35 to Week 51) were performed to evaluate long-term effects, including immunogenicity (i.e. ADAs), and the effects of repeated switching between GP2017 and Humira.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age at time of screening
* Chronic plaque-type psoriasis diagnosed for at least 6 months before randomization
* Moderate to severe psoriasis as defined at baseline by:

  * PASI score of 12 or greater
  * Investigator´s Global Assessment score of 3 or greater (based on a scale of 0 - 4) and,
  * Body Surface Area affected by plaque-type psoriasis of 10% or greater
* Chronic plaque-type psoriasis patients who have previously received phototherapy or systemic psoriasis therapy at least once or who are candidates for such therapies in the opinion of the investigator.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type
* Drug-induced psoriasis
* Ongoing use of prohibited psoriasis treatments
* Previous exposure to adalimumab
* Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of treatment with adalimumab

Other In-/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (69):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Alliance Dermatology & MOHS Center, PC, Phoenix, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Wallace Medical Group, Beverly Hills, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Dr. Howard Sofen, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Palmtree Clinical Research, Rancho Mirage, California
  - Medical Center For Clinical Research, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Ventura Clinical Trials, Ventura, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Savin Dermatology Center, P.C., New Haven, Connecticut
  - Florida Academic Dermatology Center, Coral Gables, Florida
  - Florida Medical Center & Research Inc, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Psoriasis Treatment Center of South Florida, Pembroke Pines, Florida
  - McIlwain Medical Group, PA, Tampa, Florida
  - MedPhase, Inc., Newnan, Georgia
  - Pharmaceutical Research Organization, Rigby, Idaho
  - Dundee Derm., West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Dermatology Center, PSC, New Albany, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - DermResearch, PLLC, Louisville, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Medical Development Centers, LLC, Baton Rouge, Louisiana
  - Dermat. & Adv. Aesthetics, Lake Charles, Louisiana
  - Clinical Trials of America, Inc., Monroe, Louisiana
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Associated Skin Care Specs, Fridley, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Central Dermatology, St Louis, Missouri
  - The Clinical Research Center, L.L.C., St Louis, Missouri
  - J. Woodson Dermatology & Associates, Henderson, Nevada
  - Las Vegas Skin and Cancer Clinic, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Buffalo Medical Group, P.C., Buffalo, New York
  - Forest Hills Dermatology Group, Forest Hills, New York
  - New York University Medical, Lake Success, New York
  - DermResearch Center of New York, Stony Brook, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Corvallis Clinic PC, Corvallis, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, P.C., Portland, Oregon
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Radiant Research, Inc., Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Austin Dermatology Associates, Austin, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Modern Research Associates, Dallas, Texas
  - Stephen Miller MD, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Advanced Research Institute, Ogden, Utah
  - Premier Clinical Research, Spokane, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Bulgaria (4):
  - UMHAT Dr. Georgi Stranski, EAD, Pleven
  - Center for Skin and Venereal Diseases EOOD Sofia, Sofia
  - UMHAT "Alexandrovska", EAD, Sofia
  - Diagnostic-consulting center 3-Varna EOOD, Varna
- France (2):
  - Hopital de l'Archet 2, Nice
  - Hôpital Charles Nicolle, Rouen
- Slovakia (4):
  - Kozne oddelenie,Nemocnica Kosice-Saca a.s.,1. sukromna nemoc, Kosice-Saca
  - Pedi-Derma s.r.o., Dermatovenerologicka ambulancia, Košice
  - SANARE s.r.o. Dermatovenerologická ambulancia, Svidník
  - SANARE s.r.o., Svidník

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lemke L, Blauvelt A, Bruckmann I, Cohen HP, Fan J, Guerrieri D, Horvat M, Poetzl J, Torella C, Wang Q, von Richter O. Comparing anti-drug antibody signal-to-noise ratios to assess immunogenicity and interchangeability in adalimumab biosimilar studies. Expert Opin Biol Ther. 2024 Dec;24(12):1375-1385. doi: 10.1080/14712598.2024.2428299. Epub 2024 Nov 19. PMID 39545451
- [Derived] Blauvelt A, Leonardi CL, Gaylis N, Jauch-Lembach J, Balfour A, Lemke L, Hachaichi S, Brueckmann I, Festini T, Wiland P. Treatment with SDZ-ADL, an Adalimumab Biosimilar, in Patients with Rheumatoid Arthritis, Psoriasis, or Psoriatic Arthritis: Results of Patient-Reported Outcome Measures from Two Phase III Studies (ADMYRA and ADACCESS). BioDrugs. 2021 Mar;35(2):229-238. doi: 10.1007/s40259-021-00470-1. Epub 2021 Mar 2. PMID 33651341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 661 patients were screened. 465 patients were randomized 1:1 into Treatment Period 1 and stratified by region (US/EU), body weight (<90/≥90 kg) and prior systemic therapy (no/any). In Treatment Period 2 patients were re-randomized 2:1 to either continue originally assigned treatment or switch treatment and were stratified by region only.
Pre-assignment Details: Screening lasted for at least 2 weeks and up to 4 weeks. Main inclusion criteria:
  * Men or women of at least 18 years
  * Chronic plaque-type psoriasis ≥ 6 months before randomization
  * Moderate to severe psoriasis :
    * PASI score ≥ 12
    * IGA score ≥3
    * BSA affected by plaque-type psoriasis ≥ 10%
  * No previous exposure to adalimumab
Groups:
- GP2017 Adalimumab; Humira ® Adalimumab: Solution for subcutaneous (s.c.) injection in pre-filled syringe. Study drug is administered on Day 1 with an intial dose of 80mg followed by 40mg every other week (eow) starting one week after initial dose for the first 17 weeks (Treatment Period 1).
- Humira ® Adalimumab Switched: Alternating treatment between GP2017/Humira ®/GP2017 subcutaneous (s.c.) injection of 40mg study drug (Treatment Period 2 / Week 17 until Week 35) followed by Humira ® subcutaneous (s.c.) injection of 40mg study drug (Extension Period / Week 35 until Week 51).
- Humira ® Adalimumab Continued: Humira ® subcutaneous (s.c.) injection of 40mg study drug from Week 17 until Week 35 (Treatment Period 2) and from Week 35 until Week 51 (Extension Period).
- GP2017 Adalimumab Switched: Alternating treatment between Humira ®/GP2017/Humira ® subcutaneous (s.c.) injection of 40mg study drug (Treatment Period 2 / Week 17 until Week 35) followed by GP2017 40mg subcutaneous (s.c.) injection of 40mg study drug (Extension Period / Week 35 until Week 51).
- GP2017 Adalimumab Continued: GP2017 subcutaneous (s.c.) injection of 40mg study drug from Week 17 until Week 35 (Treatment Period 2) and from Week 35 until Week 51 (Extension Period).
Period: TREATMENT PERIOD 1
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Started | 231 | 234 | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period) | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period) | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period) | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period)
Completed | 201 (12 patients did not proceed into Treatment Period 2) | 201 (11 patients did not proceed into Treatment Period 2) | 0 | 0 | 0 | 0
Not Completed | 30 | 33 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 8 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 11 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 4 | 0 | 0 | 0 | 0
Period: TREATMENT PERIOD 2
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Started | 0 (Treatment arm applicable for Treatment Period 1 only (patients re-randomized in Treatment Period 2)) | 0 (Treatment arm applicable for Treatment Period 1 only (patients re-randomized in Treatment Period 2)) | 63 (Patients re-randomized from "Humira ® adalimumab" treatment arm in Treatment Period 1) | 127 (Patients re-randomized from "Humira ® adalimumab" treatment arm in Treatment Period 1) | 63 (Patients re-randomized from "GP2017 adalimumab" treatment arm in Treatment Period 1) | 126 (Patients re-randomized from "GP2017 adalimumab" treatment arm in Treatment Period 1)
Completed | 0 | 0 | 57 | 116 | 59 | 112
Not Completed | 0 | 0 | 6 | 11 | 4 | 14
Not completed — Non compliance study medication | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2 | 6 | 3 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 1 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1
Period: EXTENSION PERIOD
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Started | 0 | 0 | 52 (5 patients did not proceed from Treatment Period 2 into Extension Period) | 109 (7 patients did not proceed from Treatment Period 2 into Extension Period) | 56 (3 patients did not proceed from Treatment Period 2 into Extension Period) | 106 (6 patients did not proceed from Treatment Period 2 into Extension Period)
Completed | 0 | 0 | 47 | 104 | 50 | 100
Not Completed | 0 | 0 | 5 | 5 | 6 | 6
Not completed — New therapy for study indication | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 3 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 2 | 2
Not completed — Non-compliance with study indication | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) consists of all randomized patients to whom a study treatment was assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab | Total
Number analyzed (Participants) | 231 | 234 | 465
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 205 | 208 | 413
  >=65 years | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (14.16) | 46.9 (14.09) | 46.3 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 92 | 181
  Male | 142 | 142 | 284
Region of Enrollment [Number; unit: participants]
  United States | 188 | 190 | 378
  Europe | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: PASI 75 Response Rate at Week 16 - GP2017 Adalimumab vs Humira ® Adalimumab
Description: The primary variable was the PASI75 response rate at Week 16, defined as the proportion of patients achieving a reduction of 75% or more of the PASI score at Week 16 compared with baseline.
Time Frame: At Week 16 only
Population: The Per-protocol analysis set (PPS) consists of patients who completed the study up to Week 16 and had no major protocol deviations or additional exclusion criteria up to and including Week 16.
Measure: Number; unit: percent of participants
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 197 | 196
percent of participants | 66.8 | 65.0
Statistical Analysis 1: Comparison: GP2017 Adalimumab vs Humira ® Adalimumab; Test type: Equivalence — Adjusted response rates were estimated using a logistic regression model including treatment, body weight strata, region and prior systemic therapy. The 95% CI for the rate difference was derived based on the normal approximation and standard error computed using the delta method.To conclude equivalent efficacy, the 95% CI had to be entirely within the interval [-18%, 18%]; Risk Difference (RD) = 1.8, 95% CI 2-sided [-7.46 to 11.15], Standard Error of Mean 4.75

2. Secondary Outcome: Mean Percent Change From Baseline in PASI Score up to Week 16 (MMRM)
Description: The key secondary efficacy variable was the percentage change from baseline in PASI score at each visit up to Week 16.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage change from baseline
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 197 | 196
percentage change from baseline | -60.7 (1.54) | -61.5 (1.55)
Statistical Analysis 1: Comparison: GP2017 Adalimumab vs Humira ® Adalimumab; Test type: Equivalence — LS means, SE and 95% CI were estimated by a Mixed Model Repeated Measures (MMRM) model with treatment, visit, treatment-by-visit interaction, body weight strata, region and prior systemic therapy, as fixed factors and baseline PASI score as covariate. Therapeutic equivalence in terms of the % change from baseline in PASI score was to be determined if the 95% CI for the difference between GP2017 and Humira treatment was contained within the interval [-15%; 15%]; LS means difference = 0.8, 95% CI 2-sided [-3.15 to 4.84], Standard Error of Mean 2.03

3. Secondary Outcome: Mean ATE of Percent Change From Baseline in PASI Score up to Week 16 (ANCOVA)
Description: The key secondary efficacy variable was the average treatment effect (ATE) which is the weighted average of % change from baseline in PASI scores between Week 1 and Week 16 (weights based on the time interval between two consecutive visits).
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage change from baseline
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 197 | 196
percentage change from baseline | -59.7 (1.59) | 60.8 (1.61)
Statistical Analysis 1: Comparison: GP2017 Adalimumab vs Humira ® Adalimumab; Test type: Equivalence — LSM, SE and 95% CI were estimated using an ANCOVA model with treatment, body weight strata, region and prior systemic therapy as fixed effects and baseline PASI score as covariate. Therapeutic equivalence in terms of the % change from baseline in PASI score was to be determined if the 95% CI for the difference between GP2017 and Humira was contained within the interval [-15%; 15%]; LS means difference = 1.2, 95% CI 2-sided [-2.78 to 5.08], Standard Error of Mean 2.0

4. Secondary Outcome: PASI 50, PASI 75, PASI 90 and PASI 100 Response Rates
Description: Proportion of patients achieving PASI 50, 75, 90 and 100 at Week 17 (end of Treatment Period 1)
Time Frame: At Week 17 only
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 197 | 196
percent of participants
  % of patients achieving PASI50 at Week 17 | 93.2 | 92.8
  % of patients achieving PASI75 at Week 17 | 71.4 | 68.6
  % of patients achieving PASI90 at Week 17 | 51.6 | 44.8
  % of patients achieving PASI100 at Week 17 | 21.9 | 16.5

5. Secondary Outcome: PASI 50, PASI75, PASI 90 and PASI100 Response Rates
Description: Proportion of Patients Achieving PASI 50, 75, 90 and 100 at Week 35 (end of Treatment Period 2)
Time Frame: At Week 35 only
Measure: Number; unit: percent of participants
Groups:
- Humira ® Adalimumab Switched: Humira is administered on Day 1 with an intial dose of 80mg followed by 40mg every other week (eow) starting one week after initial dose for the first 17 weeks (Treatment Period 1). Alternating treatment between GP2017/Humira ®/GP2017 subcutaneous (s.c.) injection of 40mg study drug (Treatment Period 2 / Week 17 until Week 35).
  Humira ® subcutaneous (s.c.) injection of 40mg study drug (Extension Period / Week 35 until Week 51).
- Humira ® Adalimumab Continued: Humira is administered on Day 1 with an intial dose of 80mg followed by 40mg every other week (eow) starting one week after initial dose until Week 51.
- GP2017 Adalimumab Switched: GP2017 is administered on Day 1 with an intial dose of 80mg followed by 40mg every other week (eow) starting one week after initial dose for the first 17 weeks (Treatment Period 1). Alternating treatment between Humira ®/GP2017/Humira ® subcutaneous (s.c.) injection of 40mg study drug (Treatment Period 2 / Week 17 until Week 35).
  GP2017 40mg subcutaneous (s.c.) injection of 40mg study drug (Extension Period / Week 35 until Week 51).
- GP2017 Adalimumab Continued: GP2017 is administered on Day 1 with an intial dose of 80mg followed by 40mg every other week (eow) starting one week after initial dose until Week 51.
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 51 | 115 | 55 | 105
percent of participants
  % of patients achieving PASI50 at Week 35 | 95.9 | 96.4 | 94.1 | 96.1
  % of patients achieving PASI75 at Week 35 | 73.5 | 73.6 | 70.6 | 74.5
  % of patients achieving PASI90 at Week 35 | 53.1 | 52.7 | 62.7 | 61.8
  % of patients achieving PASI100 at Week 35 | 28.6 | 30.9 | 35.3 | 33.3

6. Secondary Outcome: PASI 50, PASI75, PASI 90 and PASI100 Response Rates
Description: Proportion of Patients Achieving PASI 50, 75, 90 and 100 at Week 51 (Entire Study)
Time Frame: At Week 51 only
Measure: Number; unit: percent of participants
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 51 | 115 | 55 | 105
percent of participants
  % of patients achieving PASI50 at Week 51 | 95.3 | 93.9 | 87.5 | 95.9
  % of patients achieving PASI75 at Week 51 | 76.7 | 79.6 | 75.0 | 84.5
  % of patients achieving PASI90 at Week 51 | 48.8 | 51.0 | 60.4 | 62.9
  % of patients achieving PASI100 at Week 51 | 25.6 | 29.6 | 31.3 | 35.1

7. Secondary Outcome: IGA Response Rate
Description: Proportion of patients achieving a score of 0 ("clear") or 1 ("almost clear") or improved by at least 2 points of the IGA scale compared to baseline at Week 17.
Time Frame: At Week 17 only
Population: as for outcome 1
Measure: Number; unit: percent of participants
Groups:
- GP2017 Adalimumab: Study arm with intervention being studied in the protocol. Adalimumab Solution for subcutaneous injection with an initial dose of 80 mg s.c. in Week 0, followed by 40 mg s.c. eow, starting at Week 1 and ending at Week 51.
  GP2017 Adalimumab
- Humira ® Adalimumab: Humira® Adalimumab as a subcutaneous injection with an initial dose of 80 mg s.c. in Week 0, followed by 40 mg s.c. eow, starting at Week 1 and ending at Week 51.
  Humira ® Adalimumab
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 197 | 196
percent of participants | 53.6 | 53.6

8. Secondary Outcome: IGA Response Rate
Description: Proportion of patients achieving a score of 0 ("clear") or 1 ("almost clear") or improved by at least 2 points of the IGA scale compared to baseline at Week 51
Time Frame: At Week 35 only
Measure: Number; unit: percent of participants
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 51 | 115 | 55 | 105
percent of participants | 59.2 | 58.2 | 58.8 | 58.8

9. Secondary Outcome: IGA Response Rate
Description: as for outcome 8
Time Frame: At Week 51 only
Measure: Number; unit: percent of participants
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 51 | 115 | 55 | 105
percent of participants | 46.5 | 55.1 | 58.3 | 59.8

10. Secondary Outcome: DLQI
Description: Proportion of patients reporting a DLQI of 0 or 1 (no effect at all on patient's life)
Time Frame: At Week 17 only
Population: as for outcome 1
Measure: Number; unit: % of patients with DLQI of 0 or 1
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 197 | 196
% of patients with DLQI of 0 or 1 | 50.5 | 48.4

11. Secondary Outcome: DLQI
Description: Proportion of patients reporting a DLQI of 0 or 1 (no effect at all on patient's life)
Time Frame: At Week 35 only
Measure: Number; unit: % of patients with DLQI of 0 or 1
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 51 | 115 | 55 | 105
% of patients with DLQI of 0 or 1 | 49.0 | 54.5 | 52.9 | 55.9

12. Secondary Outcome: DLQI
Description: Proportion of patients reporting a DLQI of 0 or 1 (no effect at all on patient's life)
Time Frame: At Week 51 only
Measure: Number; unit: % of patients with DLQI of 0 or 1
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 51 | 115 | 55 | 105
% of patients with DLQI of 0 or 1 | 48.8 | 55.6 | 54.2 | 59.8

13. Secondary Outcome: ADA Formation Against GP2017 Adalimumab and Humira® Adalimumab From Randomization Until Week 17
Description: Proportion of patients with at least one confirmed positive anti-drug antibodies (ADA) response to adalimumab from Randomization to Week 17.
  Patients with ADA positive results at baseline were excluded from subsequent results.
Time Frame: At Week 17 only
Population: The Safety analysis set (SAF) includes all patients who received at least one dose of study treatment during Treatment Period 1. Patients were analyzed according to the treatment received.
Measure: Number; unit: % patients with at least 1 ADA+ sample
Arm/Group | GP2017 Adalimumab | Humira ® Adalimumab
Number analyzed (Participants) | 231 | 234
% patients with at least 1 ADA+ sample | 36.8 | 34.1

14. Secondary Outcome: ADA Formation Against GP2017 Adalimumab and Humira® Adalimumab From Randomization Until Week 51
Description: Proportion of patients with at least one confirmed positive anti-drug antibodies (ADA) response to adalimumab from Randomization to Week 51.
  Patients with ADA positive results at baseline were excluded from subsequent results.
Time Frame: At Week 51 only
Population: as for outcome 13
Measure: Number; unit: % patients with at least 1 ADA+ sample
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
Number analyzed (Participants) | 63 | 127 | 63 | 126
% patients with at least 1 ADA+ sample | 39.3 | 45.1 | 46.7 | 35.8

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are reported from Day 1 until the end of study (Week 51)
Arm/Group | Humira ® Adalimumab Switched | Humira ® Adalimumab Continued | GP2017 Adalimumab Switched | GP2017 Adalimumab Continued
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/127 | 0/63 | 1/126
Serious Adverse Events (participants affected / at risk) | 6/63 | 10/127 | 2/63 | 4/126
Other Adverse Events (participants affected / at risk) | 40/63 | 85/127 | 47/63 | 84/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira ® Adalimumab Switched (N=63) | Humira ® Adalimumab Continued (N=127) | GP2017 Adalimumab Switched (N=63) | GP2017 Adalimumab Continued (N=126)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotizing (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominall pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira ® Adalimumab Switched (N=63) | Humira ® Adalimumab Continued (N=127) | GP2017 Adalimumab Switched (N=63) | GP2017 Adalimumab Continued (N=126)
Nasopharyngitis (Infections and infestations) | 7 (7) | 16 (17) | 8 (12) | 12 (23)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 11 (14) | 3 (3) | 12 (17)
Sinusitis (Infections and infestations) | 2 (2) | 7 (8) | 3 (3) | 11 (13)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 2 (2) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 5 (6)
Gatroenteritis viral (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 6 (6) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 4 (4) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (4) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 7 (8) | 4 (5) | 3 (3)
Injection site erythema (General disorders) | 0 (0) | 3 (3) | 5 (14) | 6 (8)
Injection site bruising (General disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 2 (2) | 2 (15) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (5) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (5) | 1 (1) | 3 (4)
Dental caries (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (6) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 7 (8) | 2 (2) | 13 (20)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 4 (6)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 1 (1) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 10 (10) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (2) | 5 (5) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
none reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.